CLINICAL TRIAL: NCT07361367
Title: A Phase 1 Study to Evaluate the Pharmacokinetics of a Tablet Formulation of ABBV-722 and the Effect of Food on Its Bioavailability in Healthy Adult Subjects
Brief Title: A Phase 1 Study of a Tablet Form of ABBV-722 Taken With and Without Food in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-432
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Period 1: Single Dose A (Experimental): Single dose will be administered under fasted conditions
  Interventions: Drug: ABBV-722
- Period 2: Single Dose A (Experimental): Single dose will be administered under fed (high-fat meal) conditions
  Interventions: Drug: ABBV-722
- Period 3: Single Dose B (Experimental): Single dose will be administered under fasted conditions
  Interventions: Drug: ABBV-722

INTERVENTIONS:
Drug: ABBV-722 — Oral Tablet

SUMMARY:
The objective of this study is to evaluate the PK of a tablet formulation of ABBV-722 under fasted conditions and the effect of food on its bioavailability after administration of single doses

ELIGIBILITY:
Inclusion Criteria:

* Laboratory values meet the criteria specified in the protocol.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* Consumption of alcohol, grapefruit products, Seville oranges, starfruit products or quinine/tonic water within the 72-hour period prior to study drug administration.
* Use of tobacco or nicotine-containing products within 90 days prior to the first dose of study drug.
* Prior exposure to ABBV-722 within 90 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ABBV-722 | Up to Day 8 of each period (Period 1 is 9 days and Periods 2 and 3 are 8 days each; 3 periods total)
  Maximum observed plasma concentration (Cmax) of ABBV-722
Time to Cmax (Tmax) of ABBV-722 | Up to Day 8 of each period (Period 1 is 9 days and Periods 2 and 3 are 8 days each; 3 periods total)
  Time to Cmax (Tmax) of ABBV-722
Terminal Phase Elimination Rate Constant (β) of ABBV-722 | Up to Day 8 of each period (Period 1 is 9 days and Periods 2 and 3 are 8 days each; 3 periods total)
  Terminal phase elimination rate constant of ABBV-722
Terminal Phase Elimination Half-Life (t1/2) of ABBV-722 | Up to Day 8 of each period (Period 1 is 9 days and Periods 2 and 3 are 8 days each; 3 periods total)
  Terminal phase elimination half-life of ABBV-722
Area Under the Plasma Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration (AUCt) of ABBV-722 | Up to Day 8 of each period (Period 1 is 9 days and Periods 2 and 3 are 8 days each; 3 periods total)
  Area under the plasma concentration-time curve from time 0 to the time of last measurable concentration (AUCt) of ABBV-722
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinite Time (AUCinf) of ABBV-722 | Up to Day 8 of each period (Period 1 is 9 days and Periods 2 and 3 are 8 days each; 3 periods total)
  Area under the plasma concentration-time curve from time 0 to infinite time (AUCinf) of ABBV-722
Number of Participants with Adverse Events (AEs) | Up to 57 Days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 279291, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-432